CLINICAL TRIAL: NCT01157507
Title: Botulinum A Toxin Intravesical Injections Versus Bladder Overdistension in the Treatment of Patients With Painful Bladder Syndrome: A Prospective Randomized Study
Brief Title: Botulinum A Toxin in the Treatment of Patients With Painful Bladder Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Of Perugia (Other)
Responsible Party: Giannantoni Antonella, University of Perugia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MA-B-PD-P
Record Dates: First submitted 2010-02-01; First posted 2010-07-07 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2009-12

CONDITIONS: Painful Bladder Syndrome (PBS)
Keywords: Botulinum A toxin; Painful Bladder Syndrome (PBS); Bladder overdistention
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Idoxuridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Botulinum A toxin (Active Comparator): Botulinum A toxin intravesical injection.
  Interventions: Drug: Intravesical injection of Botulinum A Toxin
- Bladder overdistension (Sham Comparator): Standard treatment: bladder overdistension
  Interventions: Procedure: Bladder overdistension
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravesical injection of Botulinum A Toxin — One treatment, 100 U vials diluted in 10 ml normal saline
  Other Names: Allergan
  Arms: Botulinum A toxin
Procedure: Bladder overdistension — Bladder overdistension
  Arms: Bladder overdistension
Drug: Placebo — One single injection of placebo
  Other Names: One single injection of placebo
  Arms: Placebo

SUMMARY:
Previous clinical observations showed that Botulinum A toxin (BoNT/A) has also an antinociceptive effect and can control the neuropathic pain.

In the urologic field, recent in in vitro and in in vivo studies demonstrated that the neurotoxin is able to inhibit the release of several neurotransmitters from the bladder afferent fibers and urothelium. These neurotrasmitters as SP, CGRP, ATP, NGF and Prostaglandins are involved in neurogenic inflammation. Thus, it is reasonable to hypothesize that patients with affected by painful bladder syndrome (PBS) could benefit from BoNT/A intravesically administered.

The aim of the study is to investigate the clinical and urodynamic effects of an intravesical treatment with BoNT/A in patients affected by PBS associated with increased urinary frequency, who are refractory to conventional treatments. This treatment will be compared to bladder over distention, which is considered a conventional therapy.

DETAILED DESCRIPTION:
Patients with refractory PBS will be prospectively enrolled in the study. Baseline evaluation: Clinical evaluation with visual analog scale (VAS) for pain quantification; QoL assessment with a standardized questionnaire, HAM-A and HAM-D scales for the evaluation of anxiety and depression; voiding diary with the recording of diurnal and nocturnal urinary frequency; urodynamic evaluation, 1 month before commencing the study.

Treatment: According to a computerized randomization, patients will receive: A) one single injection of BoNT/A, 100 U diluted in 10 ml normal saline into the bladder, under cystoscopic guidance, under local anesthesia ; or B) one single bladder overdistension under local anesthesia. C) one single injection of placebo (NACL 0.9 % 10 ml) under local anesthesia.

Follow up: clinical evaluation (VAS, HAM-A and HAM-D, QOL assessment, voiding diary) and urodynamics three months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* refractory bladder pain, the urgency-frequency syndrome, and sterile urine

Exclusion Criteria:

* neurological diseases
* pregnancy and concomitant use of aminoglycosides and anticoagulants

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy: reduction in pain and diurnal and nocturnal urinary frequency; improvement in QOL; improvement in HAM-A and HAM-D scores. | PAIN quantification with 3 months follow up

SECONDARY OUTCOMES:
Urodynamic assessment | 3 months follow up

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Perugia, Perugia, Perugia, Italy